CLINICAL TRIAL: NCT06793748
Title: An Adaptive Two-Part, Phase 1/2, Multi-Center, Double-Blinded, Randomized, Controlled Study of the Safety and Efficacy of Topically Applied PEP-TISSEEL in Participants With Chronic Radiation Ulcer
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of PEP-TISSEEL in Subjects With Chronic Radiation Ulcer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rion Inc. (Industry)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-00180
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Radiation Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 1 is open label, Phase 2 is controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1-PEP-TISSEEL (Experimental): Part 1(Phase1): Participants in the PEP-TISSEEL group will receive 1 topical application per week of 2 vials of PEP + 10 mL TISSEEL for 20 weeks (5 months).
  Interventions: Combination Product: PEP-TISSEEL
- Part 1(Phase1) -TISSEEL-Only (Placebo Comparator): Part 1:Participants in the TISSEEL-Only group will receive 1 topical application per week of 10 mL TISSEEL for 20 weeks (5 months).
  Interventions: Drug: TISSEEL Fibrin Sealant KIT
- Part 2 (Phase2)-PEP-TISSEEL (Experimental): Part 2: Participants in the PEP-TISSEEL group will receive 1 topical application per week of 2 vials of PEP + 10 mL TISSEEL for 20 weeks (5 months).
  Interventions: Combination Product: PEP-TISSEEL
- Part 2(Phase2)-TISSEEL-Only (Placebo Comparator): Part 2:Participants in the TISSEEL-Only group will receive 1 topical application per week of 10 mL TISSEEL for 20 weeks (5 months).
  Interventions: Drug: TISSEEL Fibrin Sealant KIT

INTERVENTIONS:
Combination Product: PEP-TISSEEL — Purified Exosome Product (PEP™) and Fibrin Sealant (TISSEEL® VH SD Kit) (Biologic) (PEP-TISSEEL)
  Arms: Part 1-PEP-TISSEEL
Drug: TISSEEL Fibrin Sealant KIT — Fibrin Sealant (TISSEEL® VH SD Kit)
  Arms: Part 1(Phase1) -TISSEEL-Only
Combination Product: PEP-TISSEEL — Purified Exosome Product (PEP™) and Fibrin Sealant (TISSEEL® VH SD Kit) (Biologic) (PEP-TISSEEL)
  Arms: Part 2 (Phase2)-PEP-TISSEEL
Drug: TISSEEL Fibrin Sealant KIT — Fibrin Sealant (TISSEEL® VH SD Kit)
  Arms: Part 2(Phase2)-TISSEEL-Only

SUMMARY:
The goal of this clinical trial is to learn if drug Purified Exosome Product (PEP™) and Fibrin Sealant (TISSEEL® VH SD Kit) (PEP-TISSEEL) works to treat chronic radiation ulcer in adults and compare it with comparator TISSEEL. It will also learn about the safety of drug PEP-TISSEEL.

ELIGIBILITY:
Inclusion Criteria:

Participants in both study parts are eligible to be included if all of the following criteria apply:

Age and Sex

1. Males and females aged ≥ 18 years at the time of signing the informed consent. Informed Consent
2. Signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

   Type of Participant and Disease Characteristics
3. Status post-radiation treatment, with radiation-induced ulcer. This includes participants with moist desquamation as well as full epidermal necrosis and superficial dermal ulcerations (this wound would otherwise be allowed to heal by secondary intention).
4. Index ulcer classified as Grade 1 to Grade 3 according to the NCI-CTCAE, Version 5.0
5. Area of index ulcer must be between 1 and 15 cm2 at screening and at randomization/baseline.
6. Have failed conservative treatments including attempts at washing and local wound care, and be seeking therapy
7. The chronic radiation ulcers are limited to cutaneous (skin) ulcers and not impacting mucosal (oral, nose, etc.) tissue. Sex and Contraceptive/Barrier Requirements
8. Must meet one of the following criteria:

   a. Female participants of non-childbearing potential defined as : i. Postmenopausal for at least 1 year (participant verbal confirmation acceptable), or surgically sterilized (i.e., hysterectomy or bilateral oophorectomy more than 3 months prior to screening); or ii. Bilateral tubal ligation more than 6 months prior to screening; or iii. Must have a negative β-hCG blood pregnancy test at screening and not be breastfeeding prior to being administered with the IP b. Male participants of non-childbearing potential are defined as those vasectomized participants whose vasectomy was performed 6 months prior to screening or those diagnosed as sterile by a physician c. Females and males of childbearing potential who practice an acceptable method of contraception defined as the use of any form of hormonal contraceptive, a barrier method with spermicide, condoms, intrauterine device, or abstinence from sexual intercourse starting at least 60 days prior to screening and continuing at least 30 days following the last treatment. Female will undergo pregnancy tests and must have a negative β-hCG blood pregnancy test at screening visit and negative urine pregnancy test at baseline visit and must not be breastfeeding prior to being administered with the IP. Other Inclusion Criteria
9. Participants must be deemed by Radiation Oncologist at or greater than 6 months status/post-treatment to be without evidence of local recurrence
10. Ability to comply with the study protocol
11. Participants must be willing to undergo all clinical investigation-related procedures and attend all required visits including all follow-up visits Exclusion Criteria

Participants in both study parts are excluded if any of the following criteria apply:

Medical Conditions

1. Study wound exhibits clinical signs and symptoms of infection at the screening visit
2. Any participant that has vascular compromise that is untreated as defined by as by defined abnormal invasive or non-invasive vascular studies
3. The index ulcer is within 2 cm of any other ulcer
4. The non-Cutaneous CRUs and ulcers impacting mucosal (oral, nose, etc.) tissue Liver Safety
5. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN) Prior/Concurrent Clinical Study Experience
6. Use of investigational drugs or biologics within 28 days prior to screening
7. Participation in another interventional clinical study in the past 30 days or concurrent participation in another interventional clinical study Diagnostic Assessments
8. Hemoglobin A1c (HbA1c) > 8%
9. Serum creatinine l > 2.5 mg/dL
10. Absolute neutrophil count of <500 neutrophils per mm3 over the course of enrollment
11. Positive test for HBV, HCV, HIV Other Exclusion Criteria
12. Active tanning, including the use of tanning booths, during the course of the study
13. Any participant who would be unable to safely monitor the infection status of the index ulcer at home and return for scheduled visits
14. Any participant with a life expectancy ≤ 6 months
15. Pregnancy, including a positive pregnancy test at screening, or lactation
16. Likely inability to comply with the protocol or cooperate fully with the Investigator and study site personnel
17. Known or suspected active abuse of alcohol, or non-prescription drugs
18. Participants who are incarcerated for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Part 1(Phse1): Incidence of Treatment-Emergent Adverse Events (TEAEs) and Incidence of withdrawals from the study due to TEAEs | 20 week
Part 2 (Phase2): The proportion of participants with complete wound closure during the 20 weeks of the Treatment Phase | 20 weeks
  Complete wound closure of the index ulcer is defined as 100% re-epithelialization without drainage or dressing requirements confirmed at 2 consecutive study visits 2 weeks apart

SECONDARY OUTCOMES:
Part 1(Phase1): The proportion of participants with complete wound closure during the 20 weeks of the Treatment Phase | 20 weeks
  Complete wound closure of the index ulcer is defined as 100% re-epithelialization without drainage or dressing requirements confirmed at 2 consecutive study visits 2 weeks apart
Part 2(Phase2): Wound area change (%) during the 20 weeks of the Treatment Phase | 20 weeks
Part 2(Phase2): Time to complete wound closure during the 20 weeks of the Treatment Phase | 20 weeks
Part 2(Phase2):Incidence of Treatment-Emergent Adverse Events (TEAEs) | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Walker, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States